CLINICAL TRIAL: NCT05885113
Title: Developmental Intervention for Hospitalized Newborns With Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Samantha Butler, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-P00044306
Record Dates: First submitted 2023-05-09; First posted 2023-06-01 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Cardiology; Infant Development; Development Delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: This study will be a single center, single-blinded, two-arm before-and-after trial to test the feasibility of IDC vs. SOC in newborns with CHD after newborn open-heart surgery.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): NIDCAP developmental care group receiving intervention
  Interventions: Behavioral: NIDCAP Developmental Care
- standard of care (No Intervention): NO intervention, control group, receiving standard of care

INTERVENTIONS:
Behavioral: NIDCAP Developmental Care — The intervention of Individualized Developmental Care (IDC) is designed to minimize the mismatch between the fragile infant brain's expectations and the experiences of stress and pain inherent in the hospital environment. An ICU that provides individualized, developmentally-supportive care includes a soothing environment, supports parents as their child's primary caregiver, providing continual adjustment of caregiving in support of the child's wellbeing by reading the infant's cues and providing interventions to calmness throughout caregiving, capitalizing on the infant's strengths, and providing supports toward healing, growth and learning. NIDCAP is the experimental intervention to be tested in the current study. NIDCAP is the only evidence-based, comprehensive, internationally recognized program of IDC.
  Other Names: NIDCAP; Individualized Developmental Care
  Arms: Intervention

SUMMARY:
The proposed study includes a newborn developmental intervention to improve neurodevelopmental (ND) and medical outcomes for infants with congenital heart disease (CHD) with improved parent well-being. Literature documents long-term ND disabilities for children with CHD, caused by the negative effects of the hospital environment on the developing newborn brain. The cardiac intensive care unit (CICU), while necessary to save the life of the infant with CHD, exposes infants to overwhelming stress through painful procedures, invasive lines and tubes, toxic sensory stimulation, and separation from family. The combination of these negative experiences disrupts the infant's brain maturation and subsequent neurodevelopment. Individualized developmental care (IDC) is an intervention that minimizes the mismatch between infant neurobiological needs and the harsh hospital environment, thereby diminishing the frequency and severity of adverse effects. Core components of IDC include support for parent engagement, caregiving provided in a way to reduce infant stress, providing a soothing environment and appropriately positioning to enhance musculoskeletal and motor development. Research shows that IDC improves outcomes for preterm infants with enhanced brain structure and function, cognitive skills, executive functioning, behavioral outcomes, and family satisfaction from infancy to school age. Despite all the positive evidence for IDC, my past research showed most CICUs do not implement IDC due to lack of staff education and no evidence supporting IDC in CHD.

The investigators propose the first randomized controlled trial to evaluate the efficacy of IDR as an intervention for children with CHD. The investigators hypothesize infants receiving IDC provided in the hospital, compared to those not receiving IDC, will show improved medical outcomes (including shorter hospital stay, improved oral feeding, increased growth), improved developmental competence, and increased parent coping at the time of discharge home and 3 months after discharge. With support from the Children's Heart Foundation, the investigators can demonstrate the feasibility and safety of implementing IDC in the CICU, the potential to improve the ND outcome for infants with CHD and increase parent well-being. This study would serve as the needed pilot study to request funding for a larger multicenter trial which would impact CICU care of infants with CHD and their families around the world.

DETAILED DESCRIPTION:
Neurodevelopmental (ND) disabilities are the most common, and arguably the most distressing, long-term morbidity in survivors of critical congenital heart disease (CHD).1 As mortality rates for infants with CHD have declined, the need to optimize neurological and ND outcomes in survivors has assumed ever-greater importance. A myriad of studies document that longer ICU and hospital length of stay (LOS) after newborn surgery are among the strongest independent risk factors for ND delay, even after adjusting for known complications and patient factors. Few rigorous studies, however, have thoroughly tested the efficacy of bedside interventions to improve neurodevelopmental outcomes by reducing the environmental toxicities for newborns in the Cardiac Intensive Care Unit (CICU) and other in-patient settings. Individualized Developmental Care (IDC) is an intervention that maximizes the infant neurobiological needs and minimizes the harsh hospital environment, thereby diminishing the frequency and severity of adverse effects and improves long-term developmental outcomes. Core components of IDC include support and education for the family at the bedside on how to care for an ill infant, acknowledging family as the primary caregiver, incorporation of family into hands on care and positive touch, medical caregiving that reduces infant stress and supports the infant throughout, and providing a soothing environment to promote healing, growth and learning. The Newborn Individualized Developmental Care and Assessment Program (NIDCAP)2, 3 is the only evidence-based, comprehensive, internationally recognized program of IDC. IDC in the NIDCAP model has been shown to improve outcomes for premature infants with enhanced brain structure and function, along with improved behavioral outcomes that endure beyond infancy and into school age. In addition, many NIDCAP studies report benefits for medical outcomes such as decreased length of ICU and of hospital stay, earlier oral feeding, and increased weight gain.4-11 IDC as a developmental care intervention is novel in the CHD population, i.e., it has not been routinely used or tested in newborns with CHD. There is a critical need to translate this effective intervention of IDC into policy and routine care service for all infants and children hospitalized, especially those with CHD. This study supports the recent outreach to improve the implementation of effective interventions identified as a priority of health care systems and research agencies internationally.12

The proposed study would thus be the first to test the feasibility of IDC as a hospital intervention for very high-risk newborns with CHD. In this pilot single-center, single blind, before-and-after feasibility study, the investigators will compare two types of experience, standard newborn care (SOC) and the newborn intervention of developmental care (IDC) strictly following the NIDCAP model of care in the cardiology inpatient unit. The investigators will focus on the process of implementing NIDCAP care in cardiology. Following this feasibility study, the researchers will then identify strategies to address the noted challenges and/or revise components of the intervention prior to designing a multisite study to more formally evaluate the NIDCAP intervention in cardiology. Specific aims are as follows:

Primary Aim: To describe feasibility for providing IDC for infants with CHD while inpatient in cardiology. The investigators will describe organizational/contextual factors, which influence future implementation trial methods, such as recruitment, retention, data collection procedures, implementation of study protocol, and any safety concerns.

Hypothesis 1: IDC will be feasible to implement in the CICU and the cardiology step down unit/ Acute Cardiology Care Unit (ACCU). Infants who receive the IDC intervention will show an appropriate level (score of 3.5 or higher) of developmental care at the bedside during caregiving on the measure of developmental care (NIDCAP Organizational Structures Assessment13 (OSA)) scored by a study observer blind to study group. The IDC group infants will have higher scores on the OSA measurement of developmental care at the bedside than the SOC group infants.

Hypothesis 2: It will be possible to recruit enough patients into the study over the two year time frame. The investigators will collect the number of patients eligible for the study, number approached for the study, the number consented, and those that discontinue or drop from the study, along with reasoning for why someone did not meet criteria or choose to leave the study. .

Hypothesis 3: There will be no safety concerns as reported by the Safety Event Reporting System (SERS) in connection with this NIDCAP study. The investigators will review each month the number of SERS reported in the CICU and ACCU related to the study.

Secondary Aims

1. To describe the feasibility of collecting the developmental outcome assessments in this cardiac population.

   Hypothesis 1: It will be feasible to collect the Neonatal Network Neurobehavioral Scale II (NNNS) and the Developmental Assessment of Young Children-Second Edition (DAYC-2) on this population of infants. The number of missing variables will be assessed.
2. To demonstrate sufficient differentiation of developmental care and to estimate potential effect sizes to inform the design of an adequately powered trial (using the OSA scores and parent diaries).
3. To describe feasibility of increasing parent participation at the bedside, large component of NIDCAP care, for infants with CHD while inpatient in cardiology.

Hypothesis 1: Infants in the intervention group (IDC), receiving NIDCAP care will have parents who are more engaged at the bedside with higher scores (indicated increased engagement) on the Parent Risk Evaluation and Engagement Model Instrument (PREEMI) than parents of infants receiving SOC.

Hypothesis 2: Due to the increased attention to parent infant interaction given through the NIDCAP intervention, parents in the IDC group will report more time at the bedside and more daily interaction with their child on the daily diary of care than parents in the SOC group.

Our feasibility trial will provide the first, urgently needed, proof-of-concept that IDC can be implemented in hospitalized critically ill newborns with CHD. When proven to be successful, this study will provide information vital to funding of a multicenter randomized trial further expanding the knowledge of IDC for infants with CHD.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the Cardiac Intensive Care Unit (CICU) at Boston Children's Hospital (BCH) within 3 days of birth
* diagnoses of complex CHD with need for open heart surgery within the first two weeks of life (for example: total anomalous pulmonary venous connection, transposition of the great arteries, truncus arteriosus, VSD with interrupted aortic arch)
* free from associated extracardiac anomalies that are moderate or severe
* free from previous cardiac surgery or associated cardiovascular anomalies
* GA greater than 37 weeks
* 1 and 5 minute Apgar ≥ 4
* free of known chromosomal and congenital abnormalities (e.g., Down syndrome, 22q11 deletion, Noonan syndrome, Williams syndrome)
* free from multiple congenital anomalies (e.g., CHARGE syndrome)
* mother's age ≥ 20 ≤ 45 years
* absence of reported maternal alcohol, nicotine, or illegal drug use by maternal report and medical record review
* telephone/internet access.

Exclusion Criteria:

* Patients who experience cardiac arrest, CPR, ECMO, or VAD prior to recruitment

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
NIDCAP Organizational Structures Assessment (OSA)) | up to 2 months of age
  Measure of Developmental Care in the hospital at the bedside; 0-5 with 5 being the best score.

SECONDARY OUTCOMES:
Neonatal Network Neurobehavioral Scale II (NNNS) of Young Children-Second Edition (DAYC-2) | up to 2 months of age
  infant assessment; summary scores in percentile; 10-90 percentiles are considered normative performance.
Developmental Assessment of Young Children-Second Edition (DAYC-2) | at 3 months of age
  infant assessment; standard score with 100 average and S.D. of 15.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Butler, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sood E, Berends WM, Butcher JL, Lisanti AJ, Medoff-Cooper B, Singer J, Willen E, Butler S. Developmental Care in North American Pediatric Cardiac Intensive Care Units: Survey of Current Practices. Adv Neonatal Care. 2016 Jun;16(3):211-9. doi: 10.1097/ANC.0000000000000264. PMID 27140031
- [Result] Lisanti AJ, Vittner D, Medoff-Cooper B, Fogel J, Wernovsky G, Butler S. Individualized Family-Centered Developmental Care: An Essential Model to Address the Unique Needs of Infants With Congenital Heart Disease. J Cardiovasc Nurs. 2019 Jan/Feb;34(1):85-93. doi: 10.1097/JCN.0000000000000546. PMID 30303895
- [Result] Butler SC, Sadhwani A, Stopp C, Singer J, Wypij D, Dunbar-Masterson C, Ware J, Newburger JW. Neurodevelopmental assessment of infants with congenital heart disease in the early postoperative period. Congenit Heart Dis. 2019 Mar;14(2):236-245. doi: 10.1111/chd.12686. Epub 2018 Oct 15. PMID 30324749
- [Result] Miller TA, Lisanti AJ, Witte MK, Elhoff JJ, Mahle WT, Uzark KC, Alexander N, Butler SC. A Collaborative Learning Assessment of Developmental Care Practices for Infants in the Cardiac Intensive Care Unit. J Pediatr. 2020 May;220:93-100. doi: 10.1016/j.jpeds.2020.01.043. Epub 2020 Mar 5. PMID 32147219
- [Result] Als H, Duffy FH, McAnulty GB, Rivkin MJ, Vajapeyam S, Mulkern RV, Warfield SK, Huppi PS, Butler SC, Conneman N, Fischer C, Eichenwald EC. Early experience alters brain function and structure. Pediatrics. 2004 Apr;113(4):846-57. doi: 10.1542/peds.113.4.846. PMID 15060237
- [Result] Marino BS, Lipkin PH, Newburger JW, Peacock G, Gerdes M, Gaynor JW, Mussatto KA, Uzark K, Goldberg CS, Johnson WH Jr, Li J, Smith SE, Bellinger DC, Mahle WT; American Heart Association Congenital Heart Defects Committee, Council on Cardiovascular Disease in the Young, Council on Cardiovascular Nursing, and Stroke Council. Neurodevelopmental outcomes in children with congenital heart disease: evaluation and management: a scientific statement from the American Heart Association. Circulation. 2012 Aug 28;126(9):1143-72. doi: 10.1161/CIR.0b013e318265ee8a. Epub 2012 Jul 30. PMID 22851541